CLINICAL TRIAL: NCT02257008
Title: An Open Study to Investigate the Effect of Different Boosting Agents on Pharmacokinetics of Single Doses of BILR 355 BS (Dose Steps: 5 and 12.5 mg) Dissolved in 5 mL PEG 400 After Oral Administration in Healthy Male Volunteers
Brief Title: Effect of Different Boosting Agents on Pharmacokinetics of BILR 355 BS Dissolved in Polyethylene Glycol 400 (PEG 400) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1188.6
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Nelfinavir; Atazanavir Sulfate; Ritonavir

ARMS (4):
- Single rising dose of BILR 355 BS with grapefruit juice (Experimental)
  Interventions: Drug: BILR 355 BS; Other: Grapefruit juice
- Single rising dose of BILR 355 BS with nelfinavir (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Nelfinavir
- Single dose of BILR 355 BS with atazanavir (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Atazanavir
- Single dose of BILR 355 BS with atazanavir, ritonavir (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Atazanavir; Drug: Ritonavir

INTERVENTIONS:
Drug: BILR 355 BS
Other: Grapefruit juice
  Arms: Single rising dose of BILR 355 BS with grapefruit juice
Drug: Nelfinavir
  Arms: Single rising dose of BILR 355 BS with nelfinavir
Drug: Atazanavir
  Arms: Single dose of BILR 355 BS with atazanavir; Single dose of BILR 355 BS with atazanavir, ritonavir
Drug: Ritonavir
  Arms: Single dose of BILR 355 BS with atazanavir, ritonavir

SUMMARY:
Assessment of the effect of different boosting agents on pharmacokinetics of a single dose of BILR 355 BS dissolved in PEG 400

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study were to be healthy males, range from 21 to 50 years of age and their body mass index (BMI) be within 18.5 to 29.9 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters)
* In accordance with good clinical practice (GCP) and the local legislation all volunteers had to give their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (<= two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

Following exclusion criteria are of special interest for this study:

* Erythema, exanthema and comparable skin alterations
* For the boosting agents atazanavir and atazanavir plus ritonavir, subjects with a PQ interval length in the screening ECG of > 200 ms or any higher degree of atrio-ventricular (AV) block were to be excluded

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2003-03; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of the analyte in the plasma (Cmax) | up to 120 hours after start of treatment
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 120 hours after start of treatment
Area under the concentration-time curve of the analyte in plasma at different time points (AUC) | up to 120 hours after start of treatment
Apparent terminal half-life of the analyte in plasma (t1/2) | up to 120 hours after start of treatment
Apparent clearance of the analyte in plasma after extravascular multiple dose administration (CL/F) | up to 120 hours after start of treatment
Total mean residence time of the analyte in the body (MRTtot) | up to 120 hours after start of treatment
Apparent volume of distribution of the analyte during the terminal phase λz following extravascular administration (Vz/F) | up to 120 hours after start of treatment
Renal clearance of the analyte determined over the dosing interval τ (CLR) | up to 120 hours after start of treatment
Amount of the analyte excreted into urine (Ae) | up to 72 hours after start of treatment

SECONDARY OUTCOMES:
Number of participants with clinically relevant changes in laboratory parameters | up to 10 days after start of treatment
Number of participants with clinically relevant changes in vital signs (blood pressure, pulse-, respiratory rate, body temperature) | up to 10 days after start of treatment
Number of participants with clinically relevant changes in 12-lead ECG | up to 10 days after start of treatment
Number of participants with clinically relevant changes in faecal occult blood testing | up to 10 days after start of treatment
Number of participants with adverse events | Up to 25 days
Global tolerability assessment by investigator on a 5-point scale | Up to 10 days after start of treatment
Number of participants with clinically relevant changes in neurological assessment | up to 10 days after start of treatment
  Assessment of central nervous system function including Romberg's test, heel-to-toe straight line, and finger-nose tests